CLINICAL TRIAL: NCT02471547
Title: Intravesically Heated Thermo-chemotherapy With Mitomycin-C Prior to TURBT- Prospective Controlled Study
Brief Title: Intravesically Heated Thermo-chemotherapy With Mitomycin-C Prior to TURBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Ramon, Head of Urology department, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-1760-JR-CTIL
Record Dates: First submitted 2015-05-27; First posted 2015-06-15 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Transitional Cell Carcinoma
Keywords: Recurrence
MeSH Terms: conditions — Carcinoma, Transitional Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TURBT ONLY (No Intervention): A total of 150 patients in this arm will be divided into five follow-up sub groups according to pathology reports.
  Group 1 - Primary Low risk patients Group 2 - Primary Intermediate risk patients Group 3 - Primary High risk patients Group 4 - Recurrent Intermediate risk patients Group 5 - Recurrent Intermediate risk patients
- BWT with Mitomycin-C prior TURBT (Experimental): A total of 150 patients in this arm will be divided into five follow-up sub groups according to pathology reports.
  Group 1 - Primary Low risk patients Group 2 - Primary Intermediate risk patients Group 3 - Primary High risk patients Group 4 - Recurrent Intermediate risk patients Group 5 - Recurrent Intermediate risk patients
  Interventions: Other: BWT with Mitomycin-C prior TURBT

INTERVENTIONS:
Other: BWT with Mitomycin-C prior TURBT — Participants will randomly assign, according to random computerized software, to those who receive the heated thermo-chemo therapy and those who will not. The intravesical instillation will take place up to 6 hours prior TURBT in the following matter: The "Elmedical" BWT system will introduce intravesically a 40mg of heated Mitomycin MMC, diluted in 50cc of saline at a uniform temperature (44-44.50C). The length of the procedure - 50 minutes
  Other Names: Bladder wall thermo-chemotherapy (BWT)
  Arms: BWT with Mitomycin-C prior TURBT

SUMMARY:
Transurethral Resection of Bladder Tumor (TURBT) is the initial treatment procedure for urinary bladder cancer. Recurrence rate during the first year ranges between 15-38% in case of low-intermediate disease. Current literature advocate using intravesical instillations of Mitomycin-C (MMC) immediately post TURBT in order to reduce the rate of recurrence.

During the last decade, heated intravesical instillations have emerged as additional players, in the treatment of recurrent disease. By most cases, the heated intravesical instillations are given either by microwave hyperthermia (synergo®) or by conductive heat bladder wall thermo-chemotherapy (BWT).

Previous reports suggest up to 59% reduction rate in recurrence following thermo-chemotherapy upon recurrent disease. These outstanding reduction results haven't convinced significant amount of urologists worldwide to use the intravesical instillation close after endoscopic resection as TURBT, probably due to the fear of MMC adverse effects in an operated area or the fear of complications due to perforated bladder. Preliminary results have suggested favourable outcome when MMC is used prior to TURBT [see publication]. To the investigators' knowledge no previous study has prospectively examined the effect of preliminary heated intravesical installation with BWT.

DETAILED DESCRIPTION:
Scientific hypothesis: Patients treated with preliminary intravesical installation in a timely fashion before TURBT are expected to show lower recurrence rate and better outcome then control patients.

Participants: Three hundred patients designed to undergo TURBT in the urology department at "Sheba" Medical Center at "Tel Hashomer", Israel.

Exiting the research:

1. Patient is not completing the procedure due to allergic reaction or serious adverse effect during the heated intravesical instillation .
2. Patient having according to pathology report muscle invasive bladder cancer (MIBC) and expects to undergo cystectomy.

Protocol steps Eligible patients give their consent to participate in the study. A preliminary grouping (for low, intermediate and high risk groups) will be initiated according to cystoscopy examination results. (this step is for administrative purpose in order to achieve equal amount of participants between groups during follow-up phase) Then participants will randomly assign, according to randomized computer software to two major arms, those who receive the heated thermo-chemo therapy and those who will not. The intravesical instillation will take place up to 6 hours prior TURBT in the following matter: The "Elmedical" system will introduce intravesically a 40mg of heated Mitomycin-C (MMC), diluted in 50cc of saline at a uniform temperature (44-44.50C). The length of the procedure - 50 minutes.

Once pathological reports will arrive, the participant will assign to his/her actual risk group stratification. Participants with recurrent disease will be assigned into separated intermediate or high risk groups accordingly.

consequently five stratification groups are created in each major research arm (with or without prior heated intravesical instillation) Follow-up of each participant, at any group takes two years. During the follow-up period a urine cytology and routine cystoscopy will be carried out every 3 month. Patients with intermediate to high risk disease will receive six courses of intravesical bacillus Calmette-Guerin (BCG) installation according to international guidelines. Participants who for any reason won't be able to complete the BCG intravesical instillations will be offered a MMC instillation instead. Participant that pathological report is indicating a muscle invasive disease will be offered a cystectomy and exit the study (unless the participant avoids cystectomy by his/her own decision).

The investigators are obligate ourselves for surveillance according to international guidelines (as intravesical instillations of BCG or performing repeat TURBT / Biopsy by need).

Potential bias: Different surgical skills between urologists, Quality of pre-TURBT installation of thermo-chemotherapy.

Duration: Four years with two years follow up per participant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 yrs.) with good performance status according to Eastern Cooperative Oncology Group (ECOG) scale, designed to TURBT and gave their consent to participate in our research.
2. All participants must have adequate blood tests (CBC, Creatinine, electrolytes and liver function tests).

Exclusion Criteria:

1. Concurrent other malignancy in the urinary system (e.g. upper tract UC)
2. Urothelial malignancy of the bladder other then carcinoma
3. Diffuse carcinoma in situ on preliminary cystoscopy
4. Allergy or sensitivity to MMC
5. Known urinary bladder capacity of less then 200cc
6. Concurrent complicated urinary infection
7. Autoimmune disease or patient under immunosuppressive therapy
8. presence of urethral stricture
9. Previous pelvic radiotherapy
10. Concomitant malignancy of other organ
11. Pregnancy
12. Children under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of Urothelial carcinoma (UC) of bladder | Two years
  Reduced recurrence rate of Urothelial carcinoma (UC) of bladder among patients receiving intravesical heated installations

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Ramon, Prof., Principal Investigator — Sheba Medical Center, Department od Urology
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Di Stasi SM, Valenti M, Verri C, Liberati E, Giurioli A, Leprini G, Masedu F, Ricci AR, Micali F, Vespasiani G. Electromotive instillation of mitomycin immediately before transurethral resection for patients with primary urothelial non-muscle invasive bladder cancer: a randomised controlled trial. Lancet Oncol. 2011 Sep;12(9):871-9. doi: 10.1016/S1470-2045(11)70190-5. Epub 2011 Aug 8. PMID 21831711